CLINICAL TRIAL: NCT00625196
Title: A Randomised, Double-blind, Placebo-controlled, Four-way Crossover Study to Compare the Pharmacodynamics and Pharmacokinetics of GW685698X and GW642444M When Administered Separately and in Combination as a Single Dose From a Novel Dry Powder Device in Healthy Japanese Subjects
Brief Title: Comparing Two Respiratory Drugs in Combination and Separately From a Novel Inhaler Device in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: HZA102940
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Asthma
Keywords: Healthy Japanese volunteers
MeSH Terms: conditions — Asthma | interventions — vilanterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Subjects receiving fluticasone foroate/ vilanterol (Experimental): Eligible subjects will receive single dose of fluticasone foroate/ vilanterol combination treatment 800 micrograms/ 50 micrograms administered using a novel powder inhaler. There will be a washout period of 7 to 10 days between treatments.
  Interventions: Drug: Fluticasone foroate/ vilanterol; Drug: Fluticasone foroate; Drug: Vilanterol
- Subjects receiving fluticasone foroate (Active Comparator): Eligible subjects will receive single dose of fluticasone foroate 800 micrograms administered using a novel powder inhaler.
  Interventions: Drug: Fluticasone foroate
- Subjects receiving vilanterol (Active Comparator): Eligible subjects will receive single dose of vilanterol 50 micrograms administered using a novel powder inhaler.
  Interventions: Drug: Vilanterol
- Subjects receiving placebo (Placebo Comparator): Eligible subjects will receive single dose of placebo administered using a novel powder inhaler.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluticasone foroate/ vilanterol — Fluticasone foroate/ vilanterol 800 micrograms/ 50 micrograms will be available as dry powder inhaler.
  Arms: Subjects receiving fluticasone foroate/ vilanterol
Drug: Fluticasone foroate — Fluticasone foroate 800 micrograms will be available as dry powder inhaler.
  Arms: Subjects receiving fluticasone foroate; Subjects receiving fluticasone foroate/ vilanterol
Drug: Vilanterol — Vilanterol will be available as dry powder inhaler.
  Arms: Subjects receiving fluticasone foroate/ vilanterol; Subjects receiving vilanterol
Drug: Placebo — Placebo will be supplied as dry powder inhaler.
  Arms: Subjects receiving placebo

SUMMARY:
A combination of the corticosteroid GW685698X and the long-acting ß2-agonist GW642444M is being developed for once daily administration for the maintenance treatment of asthma and COPD. GW642444M and GW685698X will be simultaneously co-administered from a single device and compared with GW642444M and GW685698X administered separately in order to determine whether co-administration affects the safety, tolerability, pharmacodynamic and/or pharmacokinetics of either compound in healthy Japanese subjects.

ELIGIBILITY:
Inclusion criteria:

* Healthy male adults aged between 20 and 60 years inclusive
* Healthy as determined by a responsible physician, based on a medical evaluation including history, physical examination, laboratory tests, and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator considers that the finding will not introduce additional risk factors and will not interfere with the study procedures.
* Male subjects must use double-barrier (condom/spermicide) birth control methods or abstain from sexual intercourse with female partners who are pregnant, lactating, or able to bear children in addition to any birth control method the female partner is using, from the first dose of study medication until 90 days after the last dose of study medication.
* Japanese ethnic origin (defined as having been born in Japan with four ethnic Japanese grandparents and able to speak Japanese)
* Body weight ≥ 45 kg and body mass index within the range of 18-28 kg/m2 inclusive.
* No significant abnormality on 12-lead ECG at screening, including the following specific requirements:

  * Ventricular rate ≥ 45 beats per minute
  * PR interval ≤ 210msec
  * Q waves < 30msec (up to 50 ms permitted in lead III only)
  * QRS interval to be ≥ 60msec and ≤ 120msec
  * The waveforms must enable the QT interval to be clearly defined
  * QTc interval must be < 450msec (QTcB or QTcF; machine or manual reading) based on a single ECG value, or an average from three ECGs obtained over a brief recording period
* No significant abnormality on the Holter ECG at screening.
* FEV1 ≥90% predicted and FEV1 / FVC ratio ≥ 0.7 at screening
* Subjects who are current non- smokers who have not used any tobacco products in the 12 month period preceding the screening visit and have a pack history of < 5 pack years
* Signed and dated informed consent is obtained for the subject
* Subjects who are able to understand and comply with the protocol requirements, instructions and protocol-stated restrictions.
* Subjects who are able to use the inhalation device satisfactorily

Exclusion Criteria:

* As a result of medical interview, physical examination or screening investigations, the principle investigator or delegate physician deems the subject unsuitable for the study. Subjects must not have a systolic blood pressure above 145 mmHg or a diastolic pressure above 85 mmHg unless the Investigator confirms that it is satisfactory for their age.
* The subject has been treated for or diagnosed with depression within six months of screening or has a history of significant psychiatric illness.
* Subjects who have suffered an upper or lower respiratory tract infection within 4 weeks of the screening visit.
* Liver function tests (AST, ALT or ALP) greater than 1.5 of the upper limit of laboratory reference range.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation.
* History of milk protein allergy.
* The subject has taken prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is the longer) prior to the first dose of study medication, unless in the opinion of the Investigator and Sponsor the medication will not interfere with the study procedures or compromise subject safety.
* The subject has taken oral corticosteroids less than 8 weeks before the screening visit
* The subject has taken inhaled, intranasal or topical steroids less than 4 weeks before the screening visit
* History of alcohol/drug abuse or dependence within 12 months of the study
* Abuse of alcohol defined as an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males) or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females). One unit is equivalent to a 285mL glass of full strength beer or 425mL schooner of light beer or 1 (30mL) measure of spirits or 1 glass (100mL) of wine
* The subject has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of current study medication.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* The subject has donated a unit (450mL) of blood within the previous 16 weeks or intends to donate within 16 weeks after completing the study.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* The subject has tested positive for HIV antibodies.
* The subject has a positive pre-study urine drug screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* Positive CO or alcohol breath test at screening or on admission to the Unit.
* History of any adverse reaction including immediate or delayed hypersensitivity to any ICS, β2 agonist or sympathomimetic drug.
* Any known or suspected sensitivity to the constituents of GW642444M or GW685698X inhalation powder (i.e., lactose, magnesium stearate).
* Subjects at risk of non-compliance.

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2008-02-27 (Actual); Primary Completion 2008-05-06 (Actual); Study Completion 2008-05-06 (Actual)

PRIMARY OUTCOMES:
Maximum heart rate | over 4 hours after dosing.
Blood pressure changes | over 12 hours.
Electrocardiogram changes | over 12 hours.
Change in peak expiry flow rate changes | over 24 hours.
Change in serum cortisol concentration changes | over 24 hours

SECONDARY OUTCOMES:
Change in plasma drug concentration (AUC, Cmax, t1/2, tmax) | over 48 hours after dosing.
Change in blood potassium levels | within 4 hours of drug dosing.
Mean heart rate | over 4 hours after dosing
Plasma concentrations and derived pharmacokinetic parameters (AUC, Cmax,t½, tmax) for GW685698X, GW642444 and the GW642444 inactive metabolites GW630200 and GSK932009 | over 48 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Nakahara N, Wakamatsu A, Kempsford R, Allen A, Yamada M, Nohda S, Hirama T. The safety, pharmacokinetics and pharmacodynamics of a combination of fluticasone furoate and vilanterol in healthy Japanese subjects. Int J Clin Pharmacol Ther. 2013 Aug;51(8):660-71. doi: 10.5414/CP201822. PMID 23735179
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study HZA102940 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/HZA102940?search=study&study_ids=HZA102940#rs
- Available data/document: Informed Consent Form: HZA102940 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: HZA102940 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: HZA102940 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: HZA102940 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: HZA102940 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: HZA102940 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: HZA102940 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register